CLINICAL TRIAL: NCT00702338
Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established After Ovulation Induction in Clinical Trial 107010 for the Development of Org 36286 (Corifollitropin Alfa)
Brief Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established in Clinical Trial P05693 (P05713)
Acronym: Care
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05713; 2006-000967-26 (EudraCT Number); 107011 (Other: Organon); MK-8962-006 (Other: Merck)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Neonates
Keywords: Neonatal outcome; Congenital malformations; Ovulation Induction; Follow-up
MeSH Terms: conditions — Congenital Abnormalities | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- corifollitropin alfa + recFSH Mothers: Eligible participants in Stage 1a of base study P05693 (NCT00697255) were administered injection(s) with subcutaneous (SC) corifollitropin alfa (15mcg) and daily SC injections with recFSH (50 IU) when the largest follicle reached a size of ≥12 mm. A bolus injection of hCG (5000 IU) was then administered if at least one follicle was ≥18 mm and in total no more than two follicles ≥15 mm were observed. Eligible mothers in this group with an ongoing pregnancy established in the base study (confirmed at ≥10 weeks after hCG bolus injection) were then to be followed for safety and efficacy on the current follow-up (FU) study (P05713) according to standard practice (no treatment administered).
  Interventions: Drug: corifollitropin alfa; Biological: recombinant Follicle Stimulating Hormone (recFSH); Biological: hCG Bolus injection
- corifollitropin alfa + hCG Mothers: Eligible participants in Stage 1b of base study P05693 (NCT00697255) were administered injection(s) with SC corifollitropin alfa (30 mcg) and daily SC injections with hCG (200 IU) when the largest follicle reached a size of ≥12 mm. A bolus injection of hCG (5000 IU) was then administered if at least one follicle was ≥18 mm and in total no more than two follicles ≥15 mm were observed. Eligible mothers in this group with an ongoing pregnancy established in the base study (confirmed at ≥10 weeks after hCG bolus injection) were then followed for safety and efficacy on the current FU study (P05713) according to standard practice (no treatment administered).
  Interventions: Drug: corifollitropin alfa; Biological: human Chorion Gonadotropin (hCG); Biological: hCG Bolus injection

INTERVENTIONS:
Drug: corifollitropin alfa — SC injection(s) of corifollitropin alfa (30 mcg) was administered the first, second or third day after onset of progestagen-induced withdrawal bleeding in base study P05693 (NCT00697255). No treatment was administered on the current follow-up study.
  Other Names: Org 36286; MK-8962; SCH 900962
Biological: recombinant Follicle Stimulating Hormone (recFSH) — Daily injections of SC recFSH (50 IU/75 IU) were administered as soon as the largest follicle reached a size ≥ 12 mm 4 days after a corifollitropin alfa injection (on stimulation day 5, 9 or 13) in base study P05693 (NCT00697255). No treatment was administered on the current follow-up study.
  Groups: corifollitropin alfa + recFSH Mothers
Biological: human Chorion Gonadotropin (hCG) — Daily injections of SC hCG injection were administered as soon as the largest follicle reached a size ≥ 12 mm 4 days after a corifollitropin alfa injection (on stimulation day 5, 9 or 13) in base study P05693 (NCT00697255). No treatment was administered on the current follow-up study.
  Groups: corifollitropin alfa + hCG Mothers
Biological: hCG Bolus injection — Bolus injection of SC hCG was administered in base study P05693 (NCT00697255) to induce final oocyte maturation if at least one follicle was ≥18 mm and no more than two follicles ≥15 mm were observed. No treatment was administered on the current follow-up study.

SUMMARY:
The objective of follow-up study P05713 is to evaluate whether corifollitropin alfa (Org 36286) treatment for the induction of monofollicular growth in women who underwent ovulation induction (OI) in base study P05693 (NCT00697255) is safe for pregnant participants and their offspring.

DETAILED DESCRIPTION:
Base study P05693 (NCT00697255) was planned to include two separate stages (Ia+Ib and II).

Stage Ia was open-label and uncontrolled in a small cohort of women (n=5) to explore whether the intended dosing regimen of corifollitropin alfa followed by daily low dose recombinant Follicle Stimulating Hormone (recFSH) would provide an appropriate response in eligible participants meeting all inclusion and none of the exclusion criteria.

Stage Ib was open-label and uncontrolled in a small cohort of women (n=3) to explore whether the intended dosing regimen of corifollitropin alfa followed by daily low dose Human Chorion Gonadotropin (hCG) would provide an appropriate response in eligible participants meeting all inclusion and none of the exclusion criteria.

Stage II was planned to be open-label and randomized (n=40) to evaluate whether the intended dosing regimen of corifollitropin alfa followed by low dose recFSH (n=20) or hCG (n=20) would provide an appropriate response in eligible participants meeting all inclusion and none of the exclusion criteria.

P05713 is a follow-up (FU) study to prospectively monitor pregnancy, delivery, and neonatal outcome of women who became ongoing pregnant during base study P05693 (NCT00697255). For this trial, no study specific assessments will be required and no treatment will be administered, but information as obtained in standard practice will be used. Enrollment will begin when the first ongoing pregnancy resulting from the base study has been established (ultrasound ≥ 10 weeks after bolus injection of hCG).

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in base study P05693 (NCT00697255) and received at least one dose of corifollitropin alfa
* Ongoing pregnancy confirmed by ultrasound at least 10 weeks after bolus injection of hCG in base study P05693
* Able and willing to give written informed consent (informed consent is

incorporated in the informed consent form of protocol P05693)

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with an ongoing pregnancy at least 10 weeks after bolus injection of hCG in base study P05693 (NCT00697255).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-05-15 (Actual); Primary Completion 2008-08-09 (Actual); Study Completion 2008-12-15 (Actual)

REFERENCES:
- [Derived] Bonduelle M, Mannaerts B, Leader A, Bergh C, Passier D, Devroey P. Prospective follow-up of 838 fetuses conceived after ovarian stimulation with corifollitropin alfa: comparative and overall neonatal outcome. Hum Reprod. 2012 Jul;27(7):2177-85. doi: 10.1093/humrep/des156. Epub 2012 May 15. PMID 22587997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants treated with either corifollitropin alfa + recombinant Follicular Stimulating Hormone (recFSH) or corifollitropin alfa + Human Chorion Gonadotropin (hCG) in P05693 (NCT00697255) and with an ongoing pregnancy were to be recruited for the following study.
Pre-assignment Details: Of 8 participants treated with corifollitropin alfa + recFSH (5) or hCG (3) in base study P05693 (NCT00697255), one participant from the corifollitropin alfa + hCG group was enrolled in the current follow-up study with an ongoing multiple pregnancy. No participants from the corifollitropin alfa + recFSH group enrolled in the current follow-up study
Groups:
- Corifollitropin Alfa + hCG FU-Infants: Infants that were born to eligible mothers who received SC corifollitropin alfa plus SC hCG on base study P05693 (NCT00697255) were followed for safety and efficacy on the current follow-up study (P05713) according to standard practice.
Period: Base Study (NCT00697255)
Arm/Group | Corifollitropin Alfa + recFSH Mothers | Corifollitropin Alfa + hCG Mothers | Corifollitropin Alfa + hCG FU-Infants
Started | 5 | 3 | 0
Completed | 2 (To complete the study, participants must have received hCG bolus injection.) | 1 (To complete the study, participants must have received hCG bolus injection.) | 0
Not Completed | 3 | 2 | 0
Period: Follow-up Study: Expectant Mothers FU
Arm/Group | Corifollitropin Alfa + recFSH Mothers | Corifollitropin Alfa + hCG Mothers | Corifollitropin Alfa + hCG FU-Infants
Started | 0 (To enroll in follow-up study, confirmed pregnancy at ≥10 wks after hCG bolus injection was required) | 1 (To enroll in follow-up study, confirmed pregnancy at ≥10 wks after hCG bolus injection was required) | 0
Completed | 0 | 0 (To complete the study, participants must have completed a follow-up visit at 4-12 weeks postpartum.) | 0
Not Completed | 0 | 1 | 0
Period: Follow-up Study: Infant FU
Arm/Group | Corifollitropin Alfa + recFSH Mothers | Corifollitropin Alfa + hCG Mothers | Corifollitropin Alfa + hCG FU-Infants
Started | 0 | 0 | 2 (Participants died on day of delivery, did not complete follow-up visit at 4-12 weeks postpartum.)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of one mother with confirmed pregnancy who was treated with corifollitropin alfa + hCG in base study P05693 (NCT00697255) and enrolled in the current follow-up study. Baseline characteristics were not summarized for the infants born on study.
Arm/Group | Corifollitropin Alfa + hCG Mothers
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Mothers With ≥1 Live Born Infant During Follow-up (Take-Home Baby Rate): Protocol Defined
Description: The Take-Home Baby Rate was defined as the number of participants with an ongoing pregnancy in base study P05693 (NCT00697255) with at least one live born infant in the current follow-up study divided by the total number of participants treated in base study P05693.
Time Frame: From ≥10 weeks after bolus injection of hCG (administered in study P05693) up to time of birth on current follow-up study (up to 1 year)
Population: Intent-to-Treat group (ITT) consisted of all treated participants in base study P05693 (NCT00697255): 5 participants in Stage Ia and 3 participants in Stage Ib.
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa + recFSH Mothers | Corifollitropin Alfa + hCG Mothers
Number analyzed (Participants) | 5 | 3
percentage of participants | 0.0 | 33.3

2. Primary Outcome: Percentage of Mothers With ≥1 Live Born Infant During Follow-up (Take-Home Baby Rate): Alternate Analysis
Description: Take-Home Baby Rate was alternately defined ad hoc as the number of participants with an ongoing pregnancy in base study P05693 (NCT00697255) with at least one live born infant in the current follow-up study divided by the total number of participants who received bolus injection of hCG in the base study.
Time Frame: as for outcome 1
Population: Participants in the Intent-to-Treat group (ITT) in base study P05693 (NCT00697255) that received bolus injection of hCG.
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa + recFSH Mothers | Corifollitropin Alfa + hCG Mothers
Number analyzed (Participants) | 2 | 1
percentage of participants | 0.0 | 100.0

3. Primary Outcome: Number of Mothers With Adverse Events (AEs) During Follow-up
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From ≥10 weeks after bolus injection of hCG (administered in study P05693) up to 1 day after birth on current follow-up study (up to 1 year)
Population: Follow-up safety analysis was performed on the one expectant mother who received corifollitropin alfa + hCG on the base study P05693 (NCT00697255) and who enrolled on the follow-up study. No mothers receiving corifollitropin alfa + recFSH in the base study were enrolled in this follow-up study or included in safety analyses.
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa + recFSH Mothers | Corifollitropin Alfa + hCG Mothers
Number analyzed (Participants) | 0 | 1
participants |  | 1

4. Primary Outcome: Number of Mothers With Serious AEs (SAEs) During Follow-up
Description: An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa + recFSH Mothers | Corifollitropin Alfa + hCG Mothers
Number analyzed (Participants) | 0 | 1
participants |  | 1

5. Primary Outcome: Number of Infants With AEs During Follow-up
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From ≥10 weeks after bolus injection of hCG (administered in study P05693) up to 12 weeks after birth on current follow-up study
Population: Follow-up safety analysis was performed on the fetuses/infants delivered by the one expectant mother who received corifollitropin alfa + hCG on the base study P05693 (NCT00697255) and who enrolled on the follow-up study. There were no other eligible infants to be evaluated for safety.
Measure: Number; unit: participant
Arm/Group | Corifollitropin Alfa + hCG FU-Infants
Number analyzed (Participants) | 2
participant | 2

6. Primary Outcome: Number of Infants With SAEs During Follow-up
Description: An SAE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Corifollitropin Alfa + hCG FU-Infants: Infants that were born to eligible mothers from study P05693 (NCT00697255) were followed for safety and efficacy on the current study according to standard practice.
Arm/Group | Corifollitropin Alfa + hCG FU-Infants
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: From ≥10 weeks after bolus injection of hCG on base study P05693 (NCT00697255) up to 1 day after birth on current follow-up study (up to 1 year) for mother, planned up to 12 weeks after birth on current follow-up study for infants.
Description: Adverse events were reported for the one expectant mother who enrolled in this follow-up study and her 2 infants that were delivered on this study. No mothers receiving corifollitropin alfa + recFSH in the base study were enrolled in this follow-up study or included in safety analyses.
Arm/Group | Corifollitropin Alfa + hCG Mothers | Corifollitropin Alfa + hCG FU-Infants
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa + hCG Mothers (N=1) | Corifollitropin Alfa + hCG FU-Infants (N=2)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa + hCG Mothers (N=1) | Corifollitropin Alfa + hCG FU-Infants (N=2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in the protocol will first be submitted to the Sponsor, at least 6 weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.